CLINICAL TRIAL: NCT05076591
Title: A Phase 1, Open-Label, Multicenter, Dose Escalation Study Evaluating the Safety, Tolerability, and Preliminary Efficacy of IMM2902 in Patients with HER2-Expressing Advanced Solid Tumors
Brief Title: IMM2902, a HER2/SIRPα Bispecific MAb-Trap Antibody-receptor Fusion Protein, in Patients with HER2-expressing Advanced Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to a business decision resulting in the deprioritization of this project and with no safety concerns present, we (the trial sponsor) have decided to request the discontinuation of study IMM2902-101.
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMM2902-101
Record Dates: First submitted 2021-09-27; First posted 2021-10-13 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumor; Advanced Breast Cancer; Advanced Gastric Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IMM2902 (Experimental): IMM2902 Phase 1a Dose escalation: 0.03, 0.1, 0.25, 0.5, 1.0, 1.5, and 2.0 mg/kg through intravenous administration weekly up to 48 weeks.
  Phase 1b Dose expansion: A disease-specific dose expansion study in patients with locally advanced (unresectable) and/or metastatic breast with HER2-overexpression (Cohort 1) or HER2-low (Cohort 2), gastric/esophageal/gastroesophageal junction (GEJ) cancer with HER2-overexpression (Cohort 3) or HER2-low (Cohort 4) and other solid tumors with HER2-overexpression (Cohort 5) is aimed at further defining safety and characterizing efficacy. Dose expansion is through intravenous administration weekly up to 48 weeks.
  Interventions: Drug: IMM2902

INTERVENTIONS:
Drug: IMM2902 — a recombinant bispecific monoclonal antibody with high affinity to the dual targets, HER2 and CD47

SUMMARY:
This trial is a first-in-human, open label, multi-center, dose escalation phase 1a study followed by a disease-specific dose expansion phase 1b study to evaluate the safety, efficacy, and pharmacokinetics (PK) of IMM2902, a HER2/SIRPα bispecific mAb-Trap antibody-receptor fusion protein, in patients with HER2-expressing advanced solid tumor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Weigh greater than 30 kg
* life expectancy of at least 3 months
* Phase 1a Histologically or cytologically confirmed HER2-expressing advanced solid malignancy, who have been treated with at least one regimen of prior systemic therapy, or who refuse systemic therapy, and for which there is no curative therapy available.
* Phase 1b Histological Diagnsis There will be 5 cohorts:

Cohort 1: Histologically confirmed HER2 overexpression (HER2 IHC 3+ or HER2 IHC 2+/ISH-positive) locally advanced (unresectable) and/or metastatic breast cancer who have progression on or after at least 2 prior lines of anti-HER2 directed therapy with trastuzumab, pertuzumab, tucatinib, Fam-trastuzumab deruxtecan-nxki and T-DM1 or other anti-HER2 therapy.

Cohort 2: Histologically confirmed HER2-low (HER2 IHC 1+ or HER2 IHC 2+/ISH-negative and/or HER2 gene amplification in tumor specimen or in circulating tumor cells by ISH, NGS, or ctDNA-NGS) locally advanced (unresectable) and/or metastatic breast cancer who have progression after 2 or more lines of systemic therapy.

Cohort 3: Histologically confirmed HER2 overexpression (HER2 IHC 3+ or HER2 IHC 2+/ISH-positive) locally advanced (unresectable) and/or metastatic gastric/esophageal/gastroesophageal junction (GEJ) cancer who have progression on or after at least one prior therapy, including prior fluoropyrimidine + platinum and prior trastuzumab, and/or fam-trastuzumab deruxtecan-nxki or other prior anti-HER2 (including investigational) therapy.

Cohort 4: Histologically confirmed HER2-low (HER2 IHC 1+ or HER2 IHC 2+/ISH-negative and/or HER2 gene amplification in tumor specimen or in circulating tumor cells by ISH, NGS, or ctDNA-NGS) locally advanced (unresectable) and/or metastatic gastric/esophageal/gastroesophageal junction (GEJ) cancer who have progression after 2 or more lines of systemic therapy.

Cohort 5: Histologically confirmed HER2 overexpression (HER2 IHC 3+ or HER2 IHC 2+/ISH-positive) any other solid tumor types, including but not limited to colorectal cancer, non-small cell lung (NSCLC), ovarian cancers, that are not breast

* Has at least non-irradiated evaluable disease (target or non-target lesions) per RECIST version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Completion of prior chemotherapy systemic anticancer therapy at least 2 weeks prior to study entry.
* Radiation therapy must be completed at least 2 weeks prior to study entry. Radiated lesions may not serve as measurable disease unless they have been radiated ≥12 months prior to enrollment.
* Patients may have parenchymal brain metastases if stable (no evidence of progression) for at least 1 month after local therapy (radiation or surgery). Leptomeningeal disease is excluded.
* Patients must have adequate organ and bone marrow function within 14 days of first dose of study drug administration
* Female subject must either be of non-reproductive potential or must have a negative urine or serum prenancy test within 7 days prior to the first dose of IMM2902.

Exclusion Criteria:

* Prior anti-cancer therapy including chemotherapy, hormonal therapy, or investigational agents within 2 weeks or within at least 4 half-lives prior to IMM2902 dosing (up to a maximum of 4 weeks).
* Prior treatment with neoadjuvant or adjuvant anthracyclines within cumulative dose of doxorubicin of >400 mg/m2 or epirubicin of >800 mg/m².
* Prior treatment with CD47 or SIRPα-targeting agents.
* Trastuzumab, pertuzumab, lapatinib, tucatinib, fam-trastuzumab deruxtecan-nxki or T-DM1 within 3 weeks before first IMM2902 dosing.
* Any unresolved toxicity NCI CTCAE v5.0 Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
* Mean QT interval corrected for heart rate (QTc) ≥ 450 ms for males or QTc ≥ 470 ms for females calculated from 2 electrocardiograms (ECGs) using Fridericia's formula. Two EKGs 5 minutes (+/-2 min) apart are mandatory.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]).
* Symptomatic congestive heart failure New York Heart Association (NYHA) Function Classification II-IV, uncontrolled hypertension, acute myocardial infarction within the last 6 months, unstable angina pectoris, cardiac arrhythmia.
* Uncontrolled diabetes mellitus, Interstitial lung disease, serious gastrointestinal conditions associated with diarrhea.
* Pulmonary embolism or deep vein thrombosis within 3 months prior to the first dose of study drug.
* Uncontrolled pulmonary, renal, or hepatic dysfunction.
* Ongoing or active infection requiring systemic treatment.
* Psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints.
* Second malignancy, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, or other malignancy for which treatment was completed at least 3 years ago and for which there is no evidence of recurrence.
* Known allergic reactions to any component or excipient of IMM2902 or known allergic reactions to trastuzumab or other prior anti-HER2 (including investigational) or other monoclonal antibody ≥ Grade 3.
* Patients requiring concomitant therapeutic anticoagulation, excluding those taking low dose of anticoagulation agents for diseases such as pulmonary embolism, deep venous thrombosis.
* Known active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus.
* Known inherited or acquired bleeding disorders.
* History of hemolytic anemia or Evans syndrome, sickle cell disease, thalassemia, G6PD deficiency, hereditary spherocytosis, or hypersplenism in the last 3 months.
* Current or prior use of immunosuppressive therapy within 14 days before the first dose of IMM2902.
* Receipt of live attenuated vaccination within 30 days prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | 48 Weeks
  All toxicities will be graded according to the NCI CTCAE Version 5.0, which provides additional guidance for AEs not specifically mentioned in CTCAE. A DLTs is defined as any Grade 3 or greater AE that is assessed as related to study treatment that occurs during the 4-week DLTs observation period.
maximum tolerated dose (MTD) of IMM2902 | 48 Weeks
  Toxicity will be evaluated according to the NCI CTCAE Version 5.0.
dose for expansion (RDE) of IMM2902 | 48 Weeks
  Toxicity will be evaluated according to the NCI CTCAE Version 5.0.
Number of patients with Adverse Events（AEs） | 48 Weeks
  Graded according to the NCI CTCAE V5.0

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Huang, MD, Study Director — VP，Clinical Development; Frank Xiaodong Gan, Study Director — SVP, Clinical Development
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mary Crowley Cancer Research, Dallas, Texas
  - NEXT Virginia, LLC, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No